CLINICAL TRIAL: NCT04103632
Title: Screening and Diagnosing Exercise-induced Bronchoconstriction in Recreational Young Athletes (12-18 y)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Jessa Hospital (Other); Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S61602
Record Dates: First submitted 2019-08-27; First posted 2019-09-25 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Young Athletes; Biomarker; Exercise Induced Bronchoconstriction; Adolescent
Keywords: Athletes

STUDY DESIGN:
Intervention Model Description: Recreational young athletes from different sport disciplines will be tested for lung function, atopy, FeNO, exercise-induced bronchoconstriction (EIB) measured by EVH and biomarkers for EIB will be studied in blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young recreational athletes (12-18 years) (Experimental): Young recreational athletes (12-18 years) of different sport disciplines:
  * Indoor sports
  * Outdoor sports
  * Swimming
  * Winter sports
  Interventions: Diagnostic Test: EVH test

INTERVENTIONS:
Diagnostic Test: EVH test — * Spirometry
  * Skin prick test
  * Peripheral blood test
  * FeNO measurement

SUMMARY:
The purpose of this study is to validate the screening protocol to study risk factors of exercise-induced bronchoconstriction (EIB) obtained in our previous study in high-school elite athletes (NCT03587675), in recreational young athletes who perform intense physical exercise.

DETAILED DESCRIPTION:
Background: Physical exercise, though absolutely beneficial for human well-being, is a well-known trigger to induce bronchoconstriction. Exercise can provoke bronchoconstriction in subjects with pre-existing asthma but can also induce bronchoconstriction in otherwise healthy subjects. The latter phenomenon is called exercise-induced bronchoconstriction (EIB). EIB is frequent in the general population and might affect between 5 and 10% of them, although population based reports are scarce. EIB is most prevalent in individuals performing endurance sport disciplines, such as long distance running, duathlon and triathlon, cycling and cross-country skiing. Due to frequent intense physical training, its incidence is higher in elite athletes compared to non-elite athletes. Its prevalence in elite athletes within these endurance sport disciplines is estimated to be up to 13%. The percentage in aquatic endurance sports was surprisingly even higher and reached 20% in the Olympic games of 2008. Besides intense physical training, environmental factors such as chlorine or cold air exposure are therefore also linked to the appearance of EIB.

It remains very difficult to screen all athletes yearly for EIB. Therefore, the goal of this study is to define risk factors and/or biomarkers that might predict EIB, already at the start of their sport career. This would allow physicians to follow their lung function parameters very closely and regularly; and, if necessary, start treatment early after the first signs of EIB.

The investigators already found that atopic individuals in a young cohort of elite athletes (12-13y) had increased risk to test positive for EIB (Fisher exact test p=0.04). However, due to the high number of subjects with a positive EIB test but negative Atopy/AQUA questionnaire, the AQUA questionnaire by itself can't be used to predict EIB (p=0.4). However, one out of five questions added by our group to this questionnaire ("Do the participant suffer from wheeze during exercise?") by itself predicted EIB with 93% specificity and 24% sensitivity. Adding a second question to this ("Has a doctor ever diagnosed the participant with an allergic condition?") increased the specificity to predict a positive EIB test to 99% but lowered sensitivity to 15% only (Jonckheere AC, J Allergy Clin Immunol, 2019). Based on the preliminary data of the slightly older cohort of also elite athletes (13-18 y), fractional exhaled nitric oxide (FeNO) levels (cut off 16 ppb) may be a useful indicator of atopic phenotypes among young elite athletes. Whether atopy is a risk factor for EIB in recreational young athletes who perform intense physical exercise has to be further studied.

Hypothesis: The investigators hypothesize that the findings in the cohort of elite athletes will be similar in the cohort of recreational athletes, performing at least 12 hours of sport a week. This means that:

* They hypothesize that questionnaires (including AQUA questionnaire) can be used to screen for EIB
* They hypothesize that atopy will be a risk factor for EIB
* They hypothesize that increased FeNO levels will be a risk factor for EIB
* They hypothesize that adding blood based biomarkers increase the predictive value of the screening protocol

Aim of the study: Therefore the aim of the study is to validate the screening protocol and diagnostic EIB test in a powered (n=500) group of recreational adolescent athletes who perform their sports at least 12h/week.

Material and method: 500 recreational athletes who perform at least 12 hours of sports a week will be recruited amongst different youth sport branches including indoor sports, outdoor sports, swimming and even winter sports. Subjects will be contacted in collaboration with their local sport doctors. Subjects from East-and West Flanders will be studied at AZ Maria Middelares in Ghent by dr J Leus, subjects from Limburg will be studied at the Jessa Hospital in Hasselt and subjects from Antwerp and Flemish-Brabant will be studied in Leuven, UZ Gasthuisberg in close collaboration with prof L Dupont, copromotor of the study.

Measurements at the visit:

* Lung function will be assessed by spirometry.
* Questionnaires, including the AQUA questionnaire
* Atopy will be assessed by skin prick test for common environmental allergens
* Fractional exhaled Nitric Oxide (FeNO) measurement
* Venous puncture (1 tube)
* Eucapnic voluntary hyperventilation (EVH) test will be used as a test for EIB (adapted for this young age).

Statistical analysis: Power analysis to study the sample size has been performed based on the previous study in first grade elite athletes. Atopy was present in 35% of the subjects and EVH test was positive in 27% of these atopic subjects and 12.5% in non-atopic subjects. Probably atopy rate was accidently higher than expected in the general population (25%) Therefore a sample size of 405 subjects would allow to predict the presence of atopy and EIB with a type I error rate of 0.05 as well as a type II error rate of 0.05 at a power of 95%. The investigators expect drop-out of 15-20% of the subjects (which is more than the investigators observed in elite athletes, but consider their willingness to adhere at a screening protocol in elite athletes to be higher than that in non-elite athletes), aiming to recruit 500 subjects.

Feasibility: FWO-TBM study budget granted

ELIGIBILITY:
Inclusion Criteria:

* Recreational athletes who perform at least 12 hours of sports a week.

Exclusion Criteria:

* Acute infection in four weeks prior the test.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 346 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Detection of exercise-induced bronchoconstriction (EIB) | Baseline
  Assessed by positive eucapnic voluntary hyperventilation (EVH test): at least 10% drop in FEV1% between 5-20' after EVH

SECONDARY OUTCOMES:
Measurement of lung function by standard spirometry: FEV1 (L) and FVC (L) | Baseline
  Determination of lung obstruction based on Tiffeneau-index: FEV1(L)/FVC(L). FVC is the volume of air that can forcibly be blown out after full inspiration. FEV1 is the volume of air that can forcibly be blown out in the first second, after full inspiration. In obstructive diseases (like asthma), the tiffeneau index is reduced (<80%).
Use of atopy to predict positive EVH test | Baseline
  Atopy will be assessed by a positive skin prick test
Use of questionnaire to predict positive EVH test | Baseline
  AQUA questionnaire + additive questions An AQUA© score ≥ 6 is proposed to predict atopy in young elite athletes. In the presence of 1 or 2 additional questions (e.g. Do you suffer from wheeze during exercise?) , the specificity to point to the risk for EIB could improve.
Use of fractional exhaled nitric oxide (FeNO) levels to predict positive EVH test | Baseline
  FeNO levels in parts per billion (PPB)
Use of blood biomarker to predict positive EVH test | Baseline
  Blood CC16 levels measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Van der Eycken S, Schelpe A, Marijsse G, Dilissen E, Troosters T, Vanbelle V, Aertgeerts S, Dupont LJ, Peers K, Bullens DM, Seys SF. Feasibility to apply eucapnic voluntary hyperventilation in young elite athletes. Respir Med. 2016 Feb;111:91-3. doi: 10.1016/j.rmed.2015.12.012. Epub 2016 Jan 4. PMID 26790574
- [Background] Bonini M, Braido F, Baiardini I, Del Giacco S, Gramiccioni C, Manara M, Tagliapietra G, Scardigno A, Sargentini V, Brozzi M, Rasi G, Bonini S. AQUA: Allergy Questionnaire for Athletes. Development and validation. Med Sci Sports Exerc. 2009 May;41(5):1034-41. doi: 10.1249/MSS.0b013e318193c663. PMID 19346984
- [Background] Jonckheere AC, Seys SF, Dilissen E, Marijsse G, Schelpe AS, Van der Eycken S, Verhalle T, Vanbelle V, Aertgeerts S, Troosters T, Peers K, Dupont LJ, Bullens DMA. AQUA(c) Questionnaire as prediction tool for atopy in young elite athletes. Pediatr Allergy Immunol. 2018 Sep;29(6):648-650. doi: 10.1111/pai.12949. Epub 2018 Jul 9. No abstract available. PMID 29908073
- [Background] Jonckheere AC, Seys S, Dilissen E, Schelpe AS, Van der Eycken S, Corthout S, Verhalle T, Goossens J, Vanbelle V, Aertgeerts S, Troosters T, Peers K, Dupont L, Bullens D. Early-onset airway damage in early-career elite athletes: A risk factor for exercise-induced bronchoconstriction. J Allergy Clin Immunol. 2019 Nov;144(5):1423-1425.e9. doi: 10.1016/j.jaci.2019.07.014. Epub 2019 Jul 26. No abstract available. PMID 31356920
- [Background] Seys SF, Hox V, Van Gerven L, Dilissen E, Marijsse G, Peeters E, Dekimpe E, Kasran A, Aertgeerts S, Troosters T, Vanbelle V, Peers K, Ceuppens JL, Hellings PW, Dupont LJ, Bullens DM. Damage-associated molecular pattern and innate cytokine release in the airways of competitive swimmers. Allergy. 2015 Feb;70(2):187-94. doi: 10.1111/all.12540. PMID 25358760